CLINICAL TRIAL: NCT04891016
Title: Toripalimab Combined With FLOT Regimen in Locally Advanced Gastric cancer-a Prospective, Open, Multi-center, Phase Ⅱ Clinical Study
Brief Title: Toripalimab Plus FLOT in Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Quanli Gao, Head of immunotherapy department, Clinical professor, Leader of immunotherapy, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH immunotherapy006
Record Dates: First submitted 2021-05-10; First posted 2021-05-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Chemotherapy; Immune Checkpoint Inhibitor; Locally Advanced Gastric Carcinoma
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): patients received FLOT regimen on day 1 and toripalimab on day 3.
  Interventions: Drug: FLOT combined with toripalimab

INTERVENTIONS:
Drug: FLOT combined with toripalimab — Patients received FLOT combined with toripalimab on Day 3 every 3 weeks, for a total of 3 cycles, followed by surgical treatment. Postoperative adjuvant therapy was determined based on pathological results: if a pathological complete response (pCR) was achieved, patients received 2 additional cycles of the neoadjuvant regimen; if pCR was not achieved, patients were given 4 cycles of SOX combined with toripalimab postoperatively.
  Other Names: FLOT plus toripalimab

SUMMARY:
Neoadjuvant chemoimmunotherapy for locally advanced gastric and gastroesophageal junction (G/GEJ) cancer is currently under investigation. Most clinical studies have simply combined chemotherapy with anti-PD-1 therapy without considering the impact of chemotherapy drugs on activated immune cells. We designed this study to explore two different treatment regimens for neoadjuvant chemotherapy in patients with locally advanced G/GEJ cancer. One group received FLOT plus toripalimab on Day 1 of each cycle, every 2 weeks for 4 cycles, followed by surgery; the other group received FLOT plus toripalimab on Day 3 of each cycle, every 3 weeks for 3 cycles, followed by surgery. A total of 69 subjects were enrolled. Preliminary statistical analysis conducted one year after the last subject was enrolled revealed no statistically significant differences in pCR and MPR between the two regimens. The median DFS for both groups has not been reached, and there is no statistically significant difference in DFS between the two groups at present. Further subgroup analysis indicated that among subjects with PD-L1 CPS ≥1, the triweekly group achieved a rate of 42.1%, compared to 29.4% in the biweekly group, with no statistically significant difference between the two groups. However, the incidence of bone marrow suppression was lower in the triweekly group than in the biweekly group. Based on the preliminary findings, we plan to conduct an expanded study and transition to a multicenter clinical trial. This study aims to further validate the efficacy of the triweekly chemoimmunotherapy in patients with PD-L1 CPS ≥1 locally advanced G/GEJ cancer.

DETAILED DESCRIPTION:
Eligible patients received FLOT combined with toripalimab on Day 3 every 3 weeks, for a total of 3 cycles, followed by surgical treatment. Postoperative adjuvant therapy was determined based on pathological results: if a pathological complete response (pCR) was achieved, patients received 2 additional cycles of the neoadjuvant regimen; if pCR was not achieved, patients were given 4 cycles of SOX combined with toripalimab postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 70 ≥ Age ≥ 18 years regardless of gender
* Gastric adenocarcinoma confirmed by pathology
* no distant metastasis and resectable or potentially resectable evaluated by general surgery experts
* ECOG PS 0-1
* clinical stage T3/4 or N+ by AJCC 8.0
* PD-L1 CPS ≥1 (IHC 22C3 pharm Dx assay (Dako))
* expected lifespan over 3 months
* Adequate organ function: 1) without growth factor and blood component support in the first 2 weeks of enrollment; 2) Cardiac function: no heart disease or coronary heart disease, grade 1-2; 3) liver function: TBIL ≤ 2ULN, AST ≤ 2.5 ULN, alt ≤ 2.5 ULNX 4 Renal function: cr ≤ 1.25ULN, liver function: TBIL ≤ 2ULN, TBIL ≤ 2.5ULN, alt ≤ 2.5ULN, 4)renal function: cr ≤ 1.25ULN.
* blood pressure normal or controlled within the normal range by antihypertensive drugs
* Diabetic patients were treated with hypoglycemic drugs to control fasting blood glucose ≤ 8mmol/L
* Patients with positive hepatitis B surface antigen need to be tested for quantitative detection of hepatitis B DNA virus. HBV DNA should be less than the upper limit of the normal test value for patients with HBV infection.
* no other serious diseases conflicting with this study
* No history of other malignant tumors
* Women of childbearing age must be tested negative for blood pregnancy test within 7 days before enrollment, and subjects of childbearing age must use appropriate contraceptive measures during the trial and within 6 months after the trial
* agreement to participate in this study and signed the informed consent form

Exclusion Criteria:

* Pregnant or lactating women
* Suffered from severe infectious diseases within 4 weeks before entering the group
* Bronchial asthma requires intermittent use of bronchodilators or medical intervention
* Due to the use of immunosuppressants before coexisting diseases and the dosage of immunosuppressants ≥ 10mg/, the oral dose of prednisone lasted for more than 2 weeks
* Clinically obvious cardio-cerebrovascular diseases, including, but not limited to, severe acute myocardial infarction, instability or severe angina pectoris, coronary artery bypass surgery, congestive heart failure, ventricular arrhythmias requiring medical intervention, left ventricular ejection fraction < 50%, stroke within 6 months
* Allergic to any experimental drug and its excipients, or have a history of severe allergy, or are contraindications to experimental drugs
* Severe mental disorders
* Abnormal coagulation function (PT > 16s, APTT > 53s, TT > 21s Fib < 1.5g/L), bleeding tendency or undergoing thrombolysis or anticoagulation therapy
* Past or present pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, severe impairment of lung function, etc.
* Unable to swallow research drugs, chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis) and intestinal obstruction affect drug use and absorption
* Have a history of immunodeficiency, including positive for HIV, or suffer from other acquired, congenital immunodeficiency diseases, or have a history of organ transplant
* Other researchers evaluate those who do not meet the criteria for admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | 6 months
  the proportion of patients with no tumor cells in the postoperative specimens

SECONDARY OUTCOMES:
rate of adverse events | 3 months
  rate of adverse events
disease-free survival | 3 years
  the rate of patients who keep from disease at three years

CONTACTS AND LOCATIONS:
Overall Officials: Quanli Gao, M.D, Principal Investigator — Department of Immunotherapy, Henan Provincial Cancer Hospital
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristics, adverse reactions, postoperative pathology
Supporting Information: Study Protocol, SAP, CSR
Time Frame: every 6 months
Access Criteria: under suitable requirement

REFERENCES:
- [Background] Voorwerk L, Slagter M, Horlings HM, Sikorska K, van de Vijver KK, de Maaker M, Nederlof I, Kluin RJC, Warren S, Ong S, Wiersma TG, Russell NS, Lalezari F, Schouten PC, Bakker NAM, Ketelaars SLC, Peters D, Lange CAH, van Werkhoven E, van Tinteren H, Mandjes IAM, Kemper I, Onderwater S, Chalabi M, Wilgenhof S, Haanen JBAG, Salgado R, de Visser KE, Sonke GS, Wessels LFA, Linn SC, Schumacher TN, Blank CU, Kok M. Immune induction strategies in metastatic triple-negative breast cancer to enhance the sensitivity to PD-1 blockade: the TONIC trial. Nat Med. 2019 Jun;25(6):920-928. doi: 10.1038/s41591-019-0432-4. Epub 2019 May 13. PMID 31086347
- [Background] Loibl S, Untch M, Burchardi N, Huober J, Sinn BV, Blohmer JU, Grischke EM, Furlanetto J, Tesch H, Hanusch C, Engels K, Rezai M, Jackisch C, Schmitt WD, von Minckwitz G, Thomalla J, Kummel S, Rautenberg B, Fasching PA, Weber K, Rhiem K, Denkert C, Schneeweiss A. A randomised phase II study investigating durvalumab in addition to an anthracycline taxane-based neoadjuvant therapy in early triple-negative breast cancer: clinical results and biomarker analysis of GeparNuevo study. Ann Oncol. 2019 Aug 1;30(8):1279-1288. doi: 10.1093/annonc/mdz158. PMID 31095287
- [Background] He X, Du Y, Wang Z, Wang X, Duan J, Wan R, Xu J, Zhang P, Wang D, Tian Y, Han J, Fei K, Bai H, Tian J, Wang J. Upfront dose-reduced chemotherapy synergizes with immunotherapy to optimize chemoimmunotherapy in squamous cell lung carcinoma. J Immunother Cancer. 2020 Oct;8(2):e000807. doi: 10.1136/jitc-2020-000807. PMID 33115941
- [Background] Shitara K, Rha SY, Wyrwicz LS, Oshima T, Karaseva N, Osipov M, Yasui H, Yabusaki H, Afanasyev S, Park YK, Al-Batran SE, Yoshikawa T, Yanez P, Dib Bartolomeo M, Lonardi S, Tabernero J, Van Cutsem E, Janjigian YY, Oh DY, Xu J, Fang X, Shih CS, Bhagia P, Bang YJ; KEYNOTE-585 investigators. Neoadjuvant and adjuvant pembrolizumab plus chemotherapy in locally advanced gastric or gastro-oesophageal cancer (KEYNOTE-585): an interim analysis of the multicentre, double-blind, randomised phase 3 study. Lancet Oncol. 2024 Feb;25(2):212-224. doi: 10.1016/S1470-2045(23)00541-7. Epub 2023 Dec 19. PMID 38134948